CLINICAL TRIAL: NCT01410331
Title: A Phase II, Randomized, Double-Blind, Placebo Controlled Dose Escalation Study to Evaluate the Safety and Efficacy of JVS-100 Administered by Direct Intramuscular Injection to Cohorts of Adults With Critical Limb Ischemia
Brief Title: Study to Evaluate the Safety and Efficacy of JVS-100 Administered to Adults With Critical Limb Ischemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Juventas Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JTCS-002
Record Dates: First submitted 2011-07-14; First posted 2011-08-05 (Estimated); Last update posted 2014-10-23 (Estimated); Status verified 2014-10

CONDITIONS: Critical Limb Ischemia
Keywords: CLI; peripheral vascular disease; PVD; PAD; SDF-1
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia; Peripheral Vascular Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Cohort 1 (Experimental): Subjects will be randomized to receive either 4 mg of JVS-100 or placebo over 8 injections.
  Interventions: Biological: JVS-100(4 mg) or placebo/8 injections
- Cohort 2 (Experimental): Subjects will be randomized to receive either 8 mg of JVS-100 or placebo over 8 injections.
  Interventions: Biological: JVS-100(8 mg) or placebo/8 injections
- Cohort 3 (Experimental): Subjects will be randomized to receive either 8 mg of JVS-100 or placebo over 16 injections.
  Interventions: Biological: JVS-100(8 mg) or placebo/16 injections
- Cohort 4 (Experimental): Subjects will be randomized to receive either 16 mg of JVS-100 or placebo over 16 injections.
  Interventions: Biological: JVS-100(16 mg) or placebo/16 injections

INTERVENTIONS:
Biological: JVS-100(4 mg) or placebo/8 injections — 4 mg of JVS-100 or placebo delivered in 8 injections
  Arms: Cohort 1
Biological: JVS-100(8 mg) or placebo/8 injections — 8 mg of JVS-100 or placebo delivered in 8 injections
  Arms: Cohort 2
Biological: JVS-100(8 mg) or placebo/16 injections — 8 mg of JVS-100 or placebo delivered in 16 injections
  Arms: Cohort 3
Biological: JVS-100(16 mg) or placebo/16 injections — 16 mg of JVS-100 or placebo delivered in 16 injections
  Arms: Cohort 4

SUMMARY:
This is a double-blind, placebo controlled study designed to evaluate the safety and efficacy of JVS-100 given to adult subjects with critical limb ischemia (CLI).

DETAILED DESCRIPTION:
48 subjects diagnosed with Rutherford Class 4-5 Critical Limb Ischemia (CLI) with non-healing ulcers and/or ischemic rest pain will be enrolled in this study designed to investigate the safety and efficacy of JVS-100. JVS-100 will be delivered by direct intramuscular injection into the limbs of study subjects. Subjects will be randomized to receive a single set of direct intramuscular injections of either JVS-100 or vehicle control and will be followed for 12 months post dosing. Safety and efficacy assessments will be collected at 3 days, 4 weeks and 3, 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Men and women 40 years of age or older
* Rutherford Category 4 or 5
* Ankle systolic pressure of 70mmHg or less, or toe pressure of 50mmHg or less
* Poor option for surgical revascularization by open or endovascular strategies
* Those diabetic subjects who are on optimal diabetes treatment, with HbA1c <8.5 %
* Subject should be on stable therapy for the treatment of CLI, including statin and antiplatelet therapy
* Subject must be willing to forgo treatment with hyperbaric oxygen, nerve stimulation, ot sympathectomy for treatment of CLI 10 days prior to 45 days following injection of study drug

Exclusion Criteria:

* Life expectancy of less than 1 year
* Previous major amputation of the leg to be treated or planned major amputation within the first month following enrollment
* Patent revascularization (within 6 weeks)in the leg to be treated prior to enrollment
* NYHA Class IV heart failure
* Evidence of osteomyelitis or active infection
* Subjects with Buerger's Disease
* Subjects with a history of Systemic Lupus Erythematosus (SLE) flare
* Subjects with established chronic kidney (stage 5) requiring dialysis
* Uncontrolled blood pressure
* Significant hepatic disease
* Diabetic subjects with active proliferative retinopathy
* Immunodeficient states or subjects receiving chronic immunosuppressive therapy
* Any patient with a history of cancer unless 1)the cancer was limited to curable non-melanoma skin malignancies, or 2)the cancer was removed by successful tumor resection, with or without radiation or chemotherapy, 5 years or more prior to enrollment in this study without recurrence
* Pregnant or lactating women or subjects of childbearing potential not protected by an effective method of birth control
* Men unwilling to agree to barrier contraception or limit sexual activity
* Presence of any other condition that, in the opinion of the investigator, might compromise any aspect of the trial
* Acute coronary syndrome within 3 month prior to enrollment
* Previous treatment with angiogenic growth factors or with stem cell therapy within 1 year
* Participation in another clinical trial in the last 30 days
* Clinically significant elevations in PT/PTT/INR
* Non-heel wound size >20 cm2 (excluding toe gangrene) or heel wound size >10cm2 on the index limb
* History of drug or alcohol abuse in the last year

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2012-03; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
To Investigate the safety and tolerability of escalating doses of JVS-100 delivered via direct intramuscular injections to subjects with CLI. | 12 Months
  Safety assessments include tracking of AEs and SAEs and laboratory assessments

SECONDARY OUTCOMES:
To investigate the initial efficacy of escalating doses of JVS-100 delivered via direct intramuscular injections to subjects with CLI. | 6 months
  Efficacy measurements include: tracking of major/minor amputations,overall survival,Quality of Life,ulcer healing, & pressure assessments.

CONTACTS AND LOCATIONS:
Overall Officials: Melina Kibbe, MD, Principal Investigator — Northwestern University
Locations (7):
- United States (5):
  - Cardiology PC, Birmingham, Alabama
  - Northwestern Memorial Hospital/Northwestern University, Chicago, Illinois
  - Minneapolis Heart Institute Foundation, Minneapolis, Minnesota
  - Montefiore Medical Center, The Bronx, New York
  - Summa Health System, Akron, Ohio
- India (2):
  - Medanta-The Medicity, Haryāna
  - Sir Ganga Ram Hospital, New Delhi